CLINICAL TRIAL: NCT00125606
Title: Randomized Phase 3 Trial for Patients With AML in CR2 Comparing Total Body Irradiation (TBI) With 8Gy/Fludarabine to Conditioning With TBI 12Gy/Cyclophosphamide
Brief Title: Phase 3 Trial for AML Patients in CR2 Comparing 8Gy TBI /Fludarabine to Conditioning With TBI 12Gy/Cyclophosphamide
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient patient recruitement
Sponsor: University Hospital Muenster (Other)
Collaborators: Technische Universität Dresden (Other); Philipps University Marburg (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Hannover Medical School (Other); Ludwig-Maximilians - University of Munich (Other); University Hospital, Essen (Other); Johann Wolfgang Goethe University Hospital (Other); Deutsche Klinik fuer Diagnostik (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AML_CR2_allo_HSCT
Record Dates: First submitted 2005-07-26; First posted 2005-08-01 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; allogeneic HSCT; reduced intensity conditioning; randomized trail
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conditioning therapy with 12 Gy TBI / cyclophosphamide 120 (Active Comparator)
  Interventions: Procedure: conditioning for allogeneic HSCT
- conditioning therapy with 8 Gy TBI / fludarabine 120 (Experimental)
  Interventions: Procedure: conditioning for allogeneic HSCT

INTERVENTIONS:
Procedure: conditioning for allogeneic HSCT

SUMMARY:
For patients with acute myeloid leukemia (AML), allogeneic hematopoetic stem cell transplantation (HSCT) is one of the most potent treatment options currently available. In order to overcome the high risk of fatal treatment-related complications, reduced intensity and nonmyeloablative conditioning regimens for allogeneic HSCT are currently being explored in various hematological malignancies including AML. At least for allogeneic HSCT in AML, the optimal dose-intensity of preparative regimens for disease control at an acceptable rate of treatment-related lethal complications has not been determined. The investigators, therefore, evaluated reduced intensity myeloablative conditioning with 8 Gy TBI and fludarabine in AML patients considered ineligible for conventional conditioning in a phase 2 trial (data published in BLOOD by Stelljes et al., 2005). The results suggest that with 8 Gy TBI/fludarabine, conditioning related and unrelated donor transplants can be performed in AML patients in first or second complete remission (CR) with a remarkably low 2-year non relapse mortality (NRM) and satisfactory disease control. Based on these data a randomized phase 3 trial for patients with AML in CR≥2 is currently being conducted by the Cooperative German Transplant Study Group comparing TBI 8 Gy/fludarabine to conventionally dosed conditioning with TBI 12 Gy/cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML in second complete remission
* HLA-identical related (HLA * A, B, and DR) or HLA-compatible unrelated donor with maximum of one Ag mismatch
* Ages 18-60 years
* Written informed consent from the patient
* Written informed consent from the donor
* No major organ dysfunction

Exclusion Criteria:

* Cardiac failure (New York Heart Association [NYHA] grade II-IV)
* Renal failure (creatinine > 2.0 mg/dl)
* Hepatic failure (total bilirubin > 3 mg/dl)
* Severe neurological/psychiatric disorder
* Previous allogeneic HSCT
* Contra-indications for used drugs
* HIV infection
* Non-compliance to processing of personal data according to the protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2004-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
treatment related mortality

SECONDARY OUTCOMES:
event free survival
overall survival
cumulative incidence of acute and chronic graft-versus-host disease (GvHD)
activity index (ECOG)
organ function

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Stelljes, M.D., Principal Investigator — Department of Medicine/Hematology and Oncology
Locations (1):
- Department of Medicine/Hematology and Oncology, Münster, North Rhine-Westphalia, Germany